CLINICAL TRIAL: NCT05204901
Title: Using Magnetic Field Tracking to Confirm Nasogastric Tube Placement at Point of Care, A Feasibility Study
Brief Title: Using Magnetic Field Tracking to Confirm Nasogastric Tube Placement at Point of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Nanyang Technological University (Other); Woodlands Health Campus (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DSRB 2021/00435
Record Dates: First submitted 2021-12-05; First posted 2022-01-24 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Enteral and Supplement Feeds Adverse Reaction; Gastrointestinal Diseases; Esophagus Disorder
Keywords: nasogastric tube; chest X-ray; confirmation of placement; magnetic tracking
MeSH Terms: conditions — Gastrointestinal Diseases; Esophageal Diseases | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic tracking (Experimental): This is the only arm of the study. All 12 participants will undergo the insertion of the magnetic-tipped guidewire into their nasogastric tube after its correct placement is confirmed by chest X-ray.
  Interventions: Device: Insertion and withdrawal of a magnetic-tipped wire into the lumen of the nasogastric tube for tracking of its position

INTERVENTIONS:
Device: Insertion and withdrawal of a magnetic-tipped wire into the lumen of the nasogastric tube for tracking of its position — In each participant, the investigator will place sensors on two sites of the sternum and track the location of the magnet as it is inserted and withdrawn from the nasogastric tube in the patients.

SUMMARY:
This is a trial on the feasibility of magnetic tracking for the confirmation of nasogastric tube location in human patients.

DETAILED DESCRIPTION:
In order to address the clinical need for the localization of nasogastric tube (NGT) at point-of-care, Nanyang Technological University, Tan Tock Seng Hospital and Woodlands Health Campus co-developed the prototype of a medical device that consists of a guidewire attached to a gold-plated Neodymium magnet to be used with a T-shaped body-worn sensors connected to a laptop. The magnetic-tipped guidewire is compatible with 14Fr or larger Ryles tubes. The sensors are passive and are designed to fit on the patient's sternum beginning at the level of the second intercostal space or xiphisternum. These sensors can track the changes in magnetic flux density real-time as the magnetic-tipped guidewire is inserted into the lumen of an NGT. The tracking may be done during NGT insertion or before feeding if confirmation of its location is required. The changes in magnetic flux density will be used to determine the location of the magnet in relation to the sensors. The result of these computations will be displayed on the computer screen as a trajectory of the magnet's movement inside the NGT. At full insertion of the guidewire, the trajectory should correspond to the actual location of the NGT in the patient.

This device is currently not in use but the investigators have notified the Health Science Authority of Singapore for its use as a Clinical Research Material.

The investigators aim to recruit 12 adult patients from both gender (6 each) who would already have had NGT placement and confirmation of its position by CXR within 48 hours of NGT insertion. These patients may have a variety of body habitus and will be screened according to a detailed list of exclusion criteria that rules out a recent medical history of oesophageal or gastric surgery, cardiac stent, pacemaker, implantable defibrillator or ferromagnetic implants in the neck, thorax, abdomen, pelvis or spine.

The investigators plan to test the following hypotheses and safety parameters.

1. Concordance of our tracking with the trajectory of the NGT seen on chest X-ray
2. The vertical and horizontal range of tracking
3. The ability to detect a leftward deviation from the midline inferior to the xiphisternum
4. Test-retest reliability
5. Adverse events related to the magnetic-tipped guidewire or the sensors

ELIGIBILITY:
Inclusion Criteria:

- Patients from the general ward or the Otorhinolaryngology clinic of Tan Tock Seng Hospital who had an NGT inserted within the last 10 days and chest X-ray confirming its correct placement

* The NGT inserted is a Ryles tube size Fr 14 or 16
* COVID negative or not deemed to be infective as judged by the prevailing policies at the time of recruitment
* Age > or = 21 years
* BMI < 35
* Height < 1.9m
* Mentally competent for informed consent

Exclusion Criteria:

* • Radiological:

  * On chest X-ray, the length of the NGT distal to the gastroesophageal junction is less than 12cm, or the side-holes of the NGT can be visualized in the esophagus.
  * The NGT is kinked within 10cm of its tip
  * The chest X-ray is rotated such that the thorax is not oriented in the frontal plane
  * The NGT cannot be visualized in the mediastinum
  * The second intercostal space cannot be visualized on chest X-ray

    • Medically unstable:
  * Heart rate >=100 or <60
  * Systolic blood pressure >=160 or <100
  * SpO2 <92% in patients with chronic lung disease and <95% in patients without chronic lung disease
  * Temperature >= 38 degrees Celsius

    • Chest wall deformity:
  * Patients with pectus carinatum or excavatum, defined by physical examination

    • Patients with the following implants
  * Pacemaker
  * Automatic cardioverter defibrillator
  * Ferromagnetic coronary stents or heart valves
  * Ferromagnetic implants of the cranium, face, spine, sternum or ribs
  * Ferromagnetic surgical clips or implants in the head, neck, thorax, abdomen or pelvis

    • Following conditions within the last 30 days
  * Upper gastrointestinal bleeding
  * Oesophageal or gastric surgery
  * Stroke
  * Myocardial infarction
  * Aortic dissection
  * Ruptured aortic aneurysm

    * Allergy to neodymium, gold, epoxy or nitinol
    * Not able to understand English, Chinese, Malay or Tamil
    * Women whose last menstrual period commenced more than 4 weeks before recruitment unless they have a negative urinary or serum pregnancy test during their current admission.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Probability of visualising a leftward deviation of the magnetic tipped guide-wire inferior to the xiphisternum | 6 months
  The investigators will measure the rate of visualisation of a left-ward deviation of the magnet below the plane of xiphisternum in participants whose nasogastric tube deviates in such a way on chest X-ray.
Difference in the distance between the magnet and the datum with that between the nasogastric tube on chest X-ray and the datum | 6 months
  The investigators will compare difference in distance (measured in millimetres) between the path of the nasogastric tube seen on magnetic tracking with that seen on chest X-ray by comparing them against a vertical midline (datum) centred over the midpoint of the sternum.

SECONDARY OUTCOMES:
test-retest variability | 6 months
  The investigators will compare the distance between the magnet and the datum at the insertion of the guide-wire against that obtained at withdrawal in order to determine the variation in the accuracy of the tracking with repeated testing.
Adverse events related to the device | 6 months
  The investigators will record the incidence of magnet dislodgement, breakage of the guidewire, pain during insertion and withdrawal of the device, dermatitis over the chest wall in reaction to the sensors and any other unexpected adverse events caused by the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized IPD may be shared with other researchers upon reasonable request.

REFERENCES:
- [Result] Miyasaka M, Li H, Tay KV, Phee SJ. A Low-Cost, Point-of-Care Test for Confirmation of Nasogastric Tube Placement via Magnetic Field Tracking. Sensors (Basel). 2021 Jun 30;21(13):4491. doi: 10.3390/s21134491. PMID 34209176
- [Derived] Li H, Tay KV, Liu J, Ong CYG, Khoo HW, Zhou A, Miyasaka M, Phee SJ. Feasibility of a low-cost magnet tracking device in confirming nasogastric tube placement at point of care, a clinical trial. Sci Rep. 2024 Mar 25;14(1):7068. doi: 10.1038/s41598-024-57455-7. PMID 38528059